CLINICAL TRIAL: NCT01646372
Title: Does Instruction on Cognitive Aid Use Improve Performance and Retention of Skills? A Simulation Based Randomized Controlled Trial
Brief Title: Does Instruction on Cognitive Aid Use Improve Performance and Retention of Skills?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: The Academy for Innovation in Medical Education (Unknown); The Ottawa Hospital Academic Medical Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: OHRI-20120006
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Long-term Retention of Advanced Cardiac Life Support Skills
Keywords: Medical Education; Cognitive Aid; Crisis Resource Management; Advanced Cardiac Life Support; Skills Retention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Active Comparator): This group gets a simulation based ACLS refresher as treatment, but no access to cognitive aids for any of the tests.
  Interventions: Other: Standard Simulation Based ACLS Refresher Teaching
- 2nd Control Group (Active Comparator): This group receives a standard Simulation based ACLS refresher as the intervention, like the control group. No mention is made of Cognitive Aids in the teaching, but they are available during the post-test and retention post-test.
  Interventions: Other: Standard Simulation Based ACLS Refresher Teaching
- Cognitive Aid Group (Experimental): This group receives Cognitive Aid based teaching as the intervention. They also have access to cognitive aids for post-test and retention post-test
  Interventions: Other: Cognitive Aid based ACLS Refresher training

INTERVENTIONS:
Other: Standard Simulation Based ACLS Refresher Teaching — 45min-1 hour time. 15 minutes didactic review of 2010 ACLS guidelines followed by practice simulated megacodes
  Arms: 2nd Control Group; Control Group
Other: Cognitive Aid based ACLS Refresher training — 45min-1 hour time. 15 minutes didactic review of 2010 ACLS guidelines followed by simulated ACLS megacode practice focused on the use of Cognitive Aids to guide management.
  Arms: Cognitive Aid Group

SUMMARY:
The purpose of this study is to investigate whether formal instruction on the use of cognitive aids in managing a crisis will result in better longterm retention of knowledge and skills. In particular, this study examines the impact of cognitive aid teaching on the Advanced Cardiac Life Support course.

ELIGIBILITY:
Inclusion Criteria:

* Post-graduate Medical trainee in departments of Anesthesia, Emergency Medicine, Critical Care, Family Medicine, Internal Medicine
* Has taken ACLS Course at least once

Exclusion Criteria:

* Never taken ACLS Course

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2012-07; Primary Completion 2016-10-31 (Actual); Study Completion 2017-01-31 (Actual)

PRIMARY OUTCOMES:
ACLS Megacode Examination Scale Score | 6 months
  Simulated scenarios will be videotaped. These will be scored according to the ACLS megacode testing checklist by trained video raters

SECONDARY OUTCOMES:
Anesthesia Non-Technical Skills Scale (ANTS) | 6 Months
  Simulated Scenarios will be videotaped. Videos will be scored by trained raters according to the validated Anesthesia Nontechnical Skills Scale.

CONTACTS AND LOCATIONS:
Locations (1):
- The Ottawa Hospital, Ottawa, Ontario, Canada